CLINICAL TRIAL: NCT05170139
Title: The Effects of Caffeine on Physical Performance of Ice Hockey Players: A Cross-over Randomized Controlled Trial
Brief Title: The Effects of Caffeine on Physical Performance of Ice Hockey Players
Acronym: cafhoc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Alejandro Gómez Bruton, Lecturer, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Caffeinehockey
Record Dates: First submitted 2021-12-09; First posted 2021-12-27 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Caffeine; Athletic Performance
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Participants will be given a bottle with either caffeine and carbohydrates or just carbohydrates. All participants will complete ice-hockey specific athletic tests in both conditions.
Who Masked: Participant, Investigator
Masking Description: Participants will be given a bottle with either caffeine and carbohydrates or just carbohydrates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Experimental): Dietary Supplement: Caffeine supplementation Participants will ingest caffeine in liquid form (3mg/kg) with carbohydrates.
  Interventions: Dietary Supplement: Caffeine
- Control condition (Placebo Comparator): Participants will ingest a drink of carbohydrates without caffeine
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Caffeine — Participants will ingest a drink with 3mg/kg of body weight mixed with carbohydrates
  Arms: Caffeine
Dietary Supplement: Placebo drink — Participants will ingest the exact same drink without caffeine
  Arms: Control condition

SUMMARY:
To date, only one study has evaluated the effect of caffeine supplementation on athletic performance in ice hockey players finding a lack of ergogenic effect. This lack of effect is surprising as caffeine has been suggested to be an effective and safe nutritional supplement to improve physical performance in both trained and untrained individuals. Therefore, the aim of the present study is to evaluate the effect of acute caffeine ingestion (3mg/kg body mass). Thirteen elite adult ice-hockey male players will perform specific ice hockey performance tests in two separate days. On both occasions players will ingest 330 ml of water with lemon powertabs isostar® (86 kcal / 19g of carbohydrates) tablets, which will include in one of these days 3 mg/kg body mass of anhydrous caffeine. Players will perform a 35-m sprint, an agility test (Weave agility - slalom with puck), and a reaction test.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* Male
* Play in the Spanish ice hockey first division.

Exclusion Criteria:

* Participants taking drugs containing ephedrine or antibiotics.
* Having suffered a musculoskeletal injury in the 3 months prior to the tests.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
35m sprint time (Seconds) | One day (one hour post caffeine consumption)
  Time that participants take to skate 35 meters. Data will be collected with photoelectric cells
Agility test time (Seconds) | One day (one hour post caffeine consumption)
  Time that participants take to perform an agility circuit. Data will be collected with photoelectric cells
Reaction test time (seconds) | One day (one hour post caffeine consumption)
  Time that participants take to complete a reaction test circuit. Data will be collected with photoelectric cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided